CLINICAL TRIAL: NCT05280912
Title: Factors Associated With The Risk of Post Tonsillectomy Hemorrhage
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hadeer Gamal Mohamed, resident of otorhinolaryngology, Sohag University
Other Study IDs: HGMohamed
Record Dates: First submitted 2022-02-18; First posted 2022-03-15 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Bleeding Following Tonsillectomy (Disorder)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
factors associated with increase risk of post tonsillectomy hemorrhage and score of associated factors

DETAILED DESCRIPTION:
investigators review the medical records of patients who underwent tonsillectomy with or without adenoidectomy in our facility. None of the included patients had any known coagulopathy. The surgery was performed by several different surgeons, either otolaryngology residents or specialists, and using either cold or bipolar dissection. The procedures were performed under general anesthesia with orotracheal intubation. Bipolar electrocoagulation was used for hemostasis, as well as in some cases vicryl sutures. All medical records were reviewed according to age, gender, indications for tonsillectomy (tonsil hypertrophy causing upper airway obstruction, snoring or sleep apnea, chronic tonsillitis, peritonsillar abscess or suspected malignancy of the tonsils), coagulation profile [international normalized ratio (INR) and activated partial thromboplastin time values (aPTT)], type of surgery (tonsillectomy alone or adenotonsillectomy), surgical technique (cold or bipolar dissection), hemostasis method (bipolar electrocoagulation alone or electrocoagulation and sutures) and post-operative hemorrhage and its characterization. In this report, investigators will evaluate patients and collection of data to make a new scoring system that assesses patients according to several preoperative and postoperative factors to know the possibility of patients developing Post tonsillectomy hemorrhage. Post tonsillectomy hemorrhage is divided into two groups according to its severity: minimal hemorrhage that stopped spontaneously/after noninvasive treatment, and hemorrhage requiring reoperation for hemostasis revision in the operating room under general anesthesia.

Postoperative hemorrhage was defined as any bleeding requiring in hospital observation or treatment (medical, compression, cauterization under general anesthesia). Patients who did not seek medical attention (e.g., patients with blood-tinged sputum or only minor bleeding) were not included in the group with post-operative hemorrhage

ELIGIBILITY:
* Inclusion criteria : All cases complicated by post-tonsillectomy bleeding

  1. after elective or emergency tonsillectomy
  2. Primary Hge or secondary Hge
  3. regardless of age, the indication of surgery, surgical techniques
* Exclusion criteria:

  1. patient who have preoperative inherited bleeding disorder
  2. Patients who did not seek medical attention (e.g., patients with blood-tinged sputum or only minor bleeding) riteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All cases complicated by post-tonsillectomy bleeding
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
new scoring system for possibility of post tonsillectomy bleeding | after 4 weeks post tonsillectomy
  investigators give a degree to the participants based on the factors they have as age and sex and accompanying to post tonsillectomy bleeding as increase white blood cells and anemia

CONTACTS AND LOCATIONS:
Overall Officials: waleed AH mohammed, professor, Study Chair — sohag faculty of medicine; mohamed ER ahmed, doctor, Study Chair — sohag faculty of medicine; khaled G dahy, doctor, Study Chair — sohag faculty of medicine
Locations (1):
- Hadir Gamal Mohamed, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wall JJ, Tay KY. Postoperative Tonsillectomy Hemorrhage. Emerg Med Clin North Am. 2018 May;36(2):415-426. doi: 10.1016/j.emc.2017.12.009. Epub 2018 Feb 10. PMID 29622331
- See also: Related Info — https://europepmc.org/abstract/MED/10969475